CLINICAL TRIAL: NCT01918436
Title: TEAMS (Training Executive, Attention, and Motor Skills): - Intervention Program for Preschoolers With ADHD (Attention Deficit Hyperactivity Disorder). A Rct. Proof-of-Concept Study.
Brief Title: RCT, Proof of Concept Study of TEAMS (Training Executive, Attention and Motor Skills) Intervention Program
Acronym: TEAMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Holbaek Sygehus (Other)
Collaborators: Psychiatry Roskilde (Industry); University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Helle Annette Vibholm, MSc, Nurse Specialist, Msc, Nurse Specialist., Holbaek Sygehus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SJ-331; RESUS (Other Grant/Funding Number: Region Zealand Psychiatric Research Unit)
Record Dates: First submitted 2013-08-02; First posted 2013-08-07 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: ADHD; Attention Deficit Disorder With Hyperactivity
Keywords: Attention Deficit Hyperactivity Disorder; Neurocognitive training for preschool children with ADHD; Play intervention for children with ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TEAMS intervention (Experimental): Pre-school children age 3-6, from Region Zealand in Denmark, diagnosed with ADHD as primary diagnosis are offered participation in the RCT study of the TEAMS program.
  The intervention groups participate in eight weekly group sessions consisting of separate parent- and children's groups.
  In the child group, the children are introduced to games that are designed to enhance inhibitory control, working memory, attention, visuospatial abilities, planning, and motor skills. The parent group consists of psychoeducation and instructions in how to encourage playing these games with their children and how to support the child's development.
  Interventions: Behavioral: TEAMS intervention
- Control group (Active Comparator): The control groups receive the standard treatment program, outlined by the clinical guidelines of Region Zealand, Denmark.
  Interventions: Other: Control group

INTERVENTIONS:
Behavioral: TEAMS intervention — In the child group the children are introduced to games that are designed to enhance inhibitory control, working memory, attention, visuospatial abilities, planning, and motor skills. The parent group consists of psychoeducation and instructions in how to encourage playing these games with their children and how to support the child's development.
  Arms: TEAMS intervention
Other: Control group — The control groups receive the standard treatment program, outlined by the clinical guidelines of Region Zealand, Denmark.
  Arms: Control group

SUMMARY:
Background:

TEAMS (Training Executive Attention and Motor Skills) is a non-pharmacological, neurocognitive intervention program targeted preschool children with ADHD developed by Professor Jeffrey Halperin, and his team from New York University. The uniqueness of this program lies in the concept, based on stimulating neurocognitive growth through focused physical activity and play (Halperin et al.; 2011, 2012, in press).

Teams hypotheses:

TEAMS is based on the notions that:

1. The behavioural manifestations of ADHD are the result of deficient neural networks that affect a wide array of neurocognitive and behavioural processes which are not necessarily identical in all children with the disorder.
2. Neurodevelopment is sensitive to and can be positively affected by appropriate environmental influences.
3. Effective environmental stimulation will be best achieved within a social context.
4. The engagement of the child in the core activities of the treatment must be intrinsically rewarding (i.e., fun) in order to facilitate compliance of the intervention.

The initial research by Halperin et al. (2012)indicated significant improvement in ADHD severity from pre- to post-treatment, which also persisted 3 months later.

Objective: The aim of this study is, through a randomized controlled trial (RCT), to validate the TEAMS treatment program in a clinical setting in Denmark.

Method: Pre-school children age 3-6, from Region Zealand in Denmark, diagnosed with ADHD as primary diagnosis are offered participation in the RCT study of the TEAMS program. The control groups receive the standard treatment program, outlined by the clinical guidelines of Region Zealand. The intervention groups participate in eight weekly group sessions consisting of separate parent- and children's groups.

In the child group the children are introduced to games that are designed to enhance inhibitory control, working memory, attention, visuospatial abilities, planning, and motor skills. The parent group consists of psychoeducation and instructions in how to encourage playing these games with their children and how to support the child's development.

DETAILED DESCRIPTION:
Based on a calculation of strength:

Concurring to a statistically significant outcome the estimated cohort should be minimum 87 children. Based on Region Zealand's visitation history records the cohort is expected to be approximately 100-160 children.

Group size:

The number of participants in each treatment group depends in part on how many children have been recruited. Given the constraints of our setting, treatment groups generally consist of at least two, and up to five participants.

Staffing: Two group leaders and one student-assistant are present for every five participants in the playgroup.

For the primary efficiency measurements the project uses: ADHD-RS-IV (Attention Deficit Hyperactivity Disorder Rating Scale fourth edition), a scale for evaluating the severity of the ADHD symptoms, SDQ-DAN (Strengths and Difficulties Questionnaire - Danish translation) focuses upon the child's strengths and weaknesses in accordance with activity and attention, emotional problems, behavioural difficulties etc. For the secondary efficiency measurements the project uses: TCA (Treatment Compliance Assessment) (Halperin et al: in press), which establishes how much time the child spends on each TEAMS activity and television/computer games each day. Each day the parents fill out the TCA, as part of a logbook which also describes compliance with the TEAMS treatment project.

The questionnaires are continuously catalogued in a database facility (SurveyXact).

The TCA instrument is completed weekly during the 8 week TEAMS program.

ELIGIBILITY:
Inclusion Criteria:

* Children age 3-6, diagnosed with ADHD as primary diagnosis

Exclusion Criteria:

* Children of parents, who are not capable of cooperating in order to implement the program.
* Children living at residential institution or in an unstable environment outside the home.
* Children or parents, who do not speak/understand Danish Children, who are in medical treatment for ADHD.
* Children with significant disabilities due to comorbidity, such as autism, attachment disorder or mental retardation.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Estimated)
Dates: Start 2012-10; Primary Completion 2014-10 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Change in ADHD (Attention Deficit Hyperactivity Disorder) core symptoms: measured by ADHD-RS IV: 'Attention Deficit Hyperactivity Disorder- symptom rating scale (teacher and parent rated.) | 1 month, 3 months, 6 months

SECONDARY OUTCOMES:
Compliance with TEAMS program (TCA: Treatment Compliance Assessment)(parent rated) | paticipants will be followed for the duration of the 8 week intervention

OTHER OUTCOMES:
Change in Behavioural screening questionnaire SDQ-DAN (Strengths and Difficulties Questionnaires - DANISH translation)(parent and teacher rated) | 1 month, 3 months, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jesper Pedersed, MD,PH.D, Study Chair — Psychiatric Hospital Roskilde: Denmark
Locations (1):
- Boerne- og Ungdomspsykiatrisk afdeling, Region Sjaelland, Holbæk, Denmark

REFERENCES:
- [Derived] Vibholm HA, Pedersen J, Faltinsen E, Marcussen MH, Gluud C, Storebo OJ. Training, executive, attention and motor skills (TEAMS) training versus standard treatment for preschool children with attention deficit hyperactivity disorder: a randomised clinical trial. BMC Res Notes. 2018 Jun 8;11(1):366. doi: 10.1186/s13104-018-3478-3. PMID 29884212